CLINICAL TRIAL: NCT06504992
Title: Powdered Intrawound Vancomycin in Open Fractures: a Randomized Controlled Trial
Brief Title: Powdered Intrawound Vancomycin in Open Fractures Trial
Acronym: PIVOT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other)
Responsible Party: Principal Investigator, Madison Price, Doctor of Medicine, PI under Dr. Gabriel Larose, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS26510 (B2024:071)
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Open Fracture; Trauma; Infection, Surgical Site; Fractures, Open; Wound Infection; Fractures, Bone; Post-Operative Wound Infection
Keywords: open fracture; vancomycin; infection; trauma; intrawound
MeSH Terms: conditions — Fractures, Open; Wounds and Injuries; Surgical Wound Infection; Wound Infection; Fractures, Bone; Infections | interventions — Vancomycin; Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial blinded to participants and end-point assessors. Participants will be randomized to either receiving the treatment, intra-operative intrawound topical vancomycin powder on open fractures in addition to intravenous antibiotics with irrigation and debridement, or the control, intravenous antibiotics with irrigation and debridement alone.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Powdered, intrawound vancomycin 1000 mg at the time of definitive surgery for open fracture fixation in addition to the current best practice of intravenous antibiotics with irrigation and debridement
  Interventions: Drug: Vancomycin 1000 MG
- Control (No Intervention): Intravenous antibiotics with irrigation and debridement alone.

INTERVENTIONS:
Drug: Vancomycin 1000 MG — Powdered, intrawound vancomycin 1000 mg at the time of definitive surgery for open fracture fixation in addition to the current best practice of intravenous antibiotics with irrigation and debridement
  Other Names: Treatment
  Arms: Treatment

SUMMARY:
The purpose of this randomized control trial is to compare the rate of post-operative infection in patients with open fractures in upper or lower extremity long bones randomized to receive intra-operative intrawound topical vancomycin powder on their open fractures in addition to the current best practice of intravenous antibiotics with irrigation and debridement compared to intravenous antibiotics with irrigation and debridement alone during definitive operative fixation of the fracture.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the effect of intra-operative intrawound topical vancomycin powder on open fractures in addition to the current best practice of intravenous antibiotics with irrigation and debridement compared to intravenous antibiotics with irrigation and debridement alone during definitive fixation of the fracture on deep surgical site infection, defined as a post-operative surgical infection requiring return to the operating room for irrigation and debridement with or without hardware removal/revision within the first six months following surgery.

Secondary Objectives:

To evaluate the effect of intra-operative intrawound topical vancomycin powder on superficial surgical site infection, defined as a post-operative infection that required antibiotic treatment but no return to the operating room, readmissions to hospital for post-operative surgical infection (deep or superficial), and hardware failure, defined as hardware loosening, loss of fixation, hardware fracture, or hardware migration, visualized either on imaging or found intra-operatively.

To evaluate differences in microbe characteristics in cultures taken intra-operatively in the take-back irrigation and debridement surgery in patients with deep surgical site infection.

To evaluate if the effect of intra-operative intrawound topical vancomycin powder changes based on fracture and patient characteristics: upper extremity versus lower extremity, Gustilo Classification, patients with documented Methicillin-resistant Staphylococcus aureus (MRSA) colonization, and mechanism of injury.

To evaluate if certain fracture and patient characteristics: upper extremity versus lower extremity, Gustilo Classification, patients with documented Methicillin-resistant Staphylococcus aureus (MRSA) colonization, and by their mechanism of injury increases the risk of infection in both the treatment and control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at time of surgery
* Patients with an open fracture classified as Gustilo Type I to IIIc in the clavicle, humerus, radius, ulna, metacarpals, upper extremity phalanges (fingers), femur, tibia, fibula and metatarsals and lower extremity phalanges (toes).
* Open fracture treated operatively with plate(s) and screw(s) hardware fixation and intramedullary fixation (IM nail).
* Able to attend standard of care follow up for six months post-operatively

Exclusion Criteria:

* Patients with known vancomycin allergy, drug administration reaction, or other sensitivities to vancomycin.
* Patients who have already had definitive fracture fixation before enrollment in the study
* Patients with open fracture already infected at time of enrollment
* Patients with current positive blood cultures (bacteremia) at time of enrollment (current, meaning they have not received treatment and now have negative most-recent blood cultures).
* Patients who have other forms of local antibiotics that are left in place at the end of the definitive fixation surgery (e.g., antibiotic loaded cement or polymethyl methacrylate (PMMA) beads)
* Patients who do not speak English
* Patients who are currently pregnant
* Patients who are unable to provide consent and do not have a substitute decision maker able to provide consent
* Patients who will have severe difficulty with follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Deep surgical site infection | Within six months of definitive surgical orthopedic fixation
  A post-operative surgical infection requiring return to the operating room for irrigation and debridement with or without hardware removal/revision after the definitive fixation.

SECONDARY OUTCOMES:
Superficial surgical site infection | Within six months of definitive surgical orthopedic fixation
  A post-operative infection that required antibiotic treatment but no return to the operating room
Hardware failure visualized either on imaging or found intra-operatively, until six months post definitive fixation | Up until six months following definitive fixation
  Hardware loosening, loss of fixation, hardware fracture, or hardware migration visualized either on imaging or found intra-operatively
Microbe sensitivity | Up until six months following definitive fixation
  In patients with deep surgical site infection, the gram stain and sensitivity and resistance to antibiotics of cultures taken intra-operatively in the take-back irrigation and debridement surgery
Fracture location | At time of initial open fracture
  Whether the fracture is in the upper extremity: clavicle, humerus, radius, ulna, metacarpals and phalanges (fingers) versus lower extremity: femur, tibia, fibula, metatarsals, and phalanges (toes).
Fracture Gustilo Classification | At time of definitive surgical orthopedic fixation.
  Open fracture classification from Type I to IIIc that classifies open fractures based on extent of bone, soft tissue and vascular injuries.
Mechanism of injury | At time of initial open fracture
  Mechanism of injury will be categorized as:
  i. Motor vehicle collision: car occupant, pedestrian, motorcyclist, other ii. Other Vehicle Accident: all-terrain vehicle (ATV), bicycle, snowmobile iii. Fall: from own height (slip/stumble), from height less than or equal to 3 metres, from height greater than 3 metres iv. Laceration v. Striking with blunt object (unintentional) vi. Crush injury vii. Sport related injury viii. Interpersonal violence: stabbing, striking with sharp object (e.g., machete), striking with blunt object, gunshot, other
MRSA colonization | During initial admission to hospital for open fracture
  Nasal swab for MRSA that is routinely taken for all patients admitted to the study's hospital

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Larose, MD, MSc, FRCSC, Principal Investigator — University of Manitoba; Madison Price, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Winnipeg, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No